CLINICAL TRIAL: NCT07107438
Title: Effect of Digital Interactive Classroom Using Thinqi Platform on Undergraduate Critical Care Nursing Students' Knowledge Retention & Engagement.
Brief Title: Digital Interactive Classroom Effect on Nursing Students' Knowledge Retention & Engagement.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heba.Attia@nur.dmu.edu.eg (Other)
Responsible Party: Sponsor-Investigator, Heba.Attia@nur.dmu.edu.eg, Faculty member " Lecturer", Damanhour University
Organization: Damanhour University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Digital Interactive Classroom
Record Dates: First submitted 2025-07-22; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Knowledge Level; Engagement
Keywords: Thinqi platform; Knowledge retension; engagment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): The interventional group will involve 50 nursing students.
  Interventions: Other: The interventional group will be trained on ECG interpretation through thinqi digital interactive platform
- Conventional group (Placebo Comparator): The conventional group will involve 50 nursing also.
  Interventions: Other: The interventional group will be trained on ECG interpretation through thinqi digital interactive platform

INTERVENTIONS:
Other: The interventional group will be trained on ECG interpretation through thinqi digital interactive platform — The conventional group will be trained on ECG interpretation through handout exercises

SUMMARY:
The study aims to determine the effect of digital interactive classroom using thinqi platform on undergraduate critical care nursing students' knowledge retention and engagement

DETAILED DESCRIPTION:
Digital platforms are educational tools that improve learning processes and provide a set of tools that allow synchronous and asynchronous interaction and communication between students themselves on one hand, and between the teacher and his students on the other hand. They also enable participation in different tasks. Digital platforms that can be used in the educational process to provide flexible and reliable learning environment are numerous such as Blackboard, Moodle, Canvas, Edmodo, Google Classroom and Thinqi.

Thinqi is a platform with key features like course management and assignment creation. Also, it offers reports and statistics on student achievement. Furthermore, Thinqi platform is flexible, scalable, versatile of use, provides discussion forums, and allows live chat between learners and teacher and between learners themselves, also it provide interaction and cooperative tools that incorporate various multimedia elements like videos images and external links to enhance learning experiences and a digital library for storing and sharing digital learning materials.

ELIGIBILITY:
Inclusion Criteria:

* Nursing students (100) who will be registered in the second academic level and enrolled in the "Emergency Nursing Course"

Exclusion Criteria:

* Other nursing students who will be registered in other academic levels and other courses

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Undergraduate Critical Care Nursing Students' Knowledge Retention | baseline and after one month of quiz
  knowledge retention will be measured through 30 MCQs quiz and the mean will be compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Hala Eid, Assistant Professor, Principal Investigator — Assistant professor of nursing education
Locations (1):
- Faculty of Nursing, Damanhour University, Damanhūr, Egypt

IPD SHARING:
Plan to Share IPD: Yes
1AA2BB3CC4DD5EE6FF7GG
Supporting Information: Study Protocol
Time Frame: at January 2026, and will be available for 2 years
Access Criteria: any researcher will be able to access the IPD foe study protocol through contacting us
URL: https://r.search.yahoo.com/_ylt=AwrEa08v_YloGAIAkuZXNyoA;_ylu=Y29sbwNiZjEEcG9zAzEEdnRpZAMEc2VjA3Ny/RV=2/RE=1755083312/RO=10/RU=https%3a%2f%2fclinicaltrials.gov%2f/RK=2/RS=A.BGLc9DHAInknyHYP6QJWH.530-